CLINICAL TRIAL: NCT03506724
Title: Ethnic Differences in Anti-Hypertensive Medication Response Among Pregnant and Postpartum Patients
Brief Title: Response to Anti-hypertensives in Pregnant and Postpartum Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Mount Sinai Hospital, New York (Other); Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Dyese Taylor, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0257; Maimonides IRB 2018-02-17 (Other: Maimonides IRB/Research Committee)
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hypertension in Pregnancy; Preeclampsia
Keywords: Hypertension, Pregnancy-induced; Pregnancy Induced Hypertension; Gestational Hypertension; Transient Hypertension, Pregnancy; Pharmacogenetics
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Nifedipine; Labetalol

STUDY DESIGN:
Intervention Model Description: Patients who present to the hospitals in this study will be randomized to receive IV labetalol or oral nifedipine when presenting with persistent severe range blood pressures (2 readings or more within 15 minutes) of either 160mmHg systolic or 110mmHg diastolic. These anti-hypertensives are first line therapy for management of severe range blood pressures by the American Congress of Obstetricians and Gynecologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral nifedipine (Other): Oral medication 10mg and 20mg
  Interventions: Drug: Nifedipine
- Intravenous labetalol (Other): intravenous medication 20mg, 40mg, 80 mg
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Nifedipine — Nifedipine 10mg oral will be given and the MAP will then be calculated 20 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, nifedipine 20mg oral will be given and the MAP will then be calculated 20 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, nifedipine 20mg oral will be given and the MAP will then be calculated 20 minutes after medication is given and institution specific protocol will be performed.
  Arms: Oral nifedipine
Drug: Labetalol — Labetalol 20mg IV will be given over 2 minutes and the MAP will then be calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, labetalol 40mg IV will be given over 2 minutes and the MAP will then be calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, labetalol 80mg IV will be given over 2 minutes and the MAP will then be calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, then another medication will be chosen based on institution specific protocol.
  Arms: Intravenous labetalol

SUMMARY:
In this study, the investigators will evaluate the blood pressure response to nifedipine and labetalol in pregnant and postpartum patients, who present with hypertensive disease in pregnancy with severe range blood pressure defined as greater than 160/110. These anti-hypertensives are first line therapy for management of severe range blood pressures in pregnancy and postpartum by the American Congress of Obstetricians and Gynecologist (ACOG). In addition at the Mount Sinai West site, the investigators will also analyze the ADRB1 and similar genes involved in beta blockade, genes involved in calcium channel blockade and other genes implicated in blood pressure response among pregnant and postpartum patients receiving labetalol and nifedipine. This analysis will be used to determine if a pharmacogenetic association exists between variant alleles in these receptors in the pregnant and postpartum population.

DETAILED DESCRIPTION:
Hypertensive disease in pregnancy is a major cause of maternal morbidity and mortality. This condition is responsible for about 12% of the maternal deaths in the United States.

Currently, if pregnant patients present with severe hypertension they are either given IV labetalol, IV hydralazine of nifedipine based on individual provider preference. There are few studies in the literature comparing oral nifedipine and IV labetalol with mixed data showing either they are equally effective or a faster time to achieving target blood pressure for patients who received nifedipine.

In this study, the investigators will evaluate if there is a difference in time to achieve goal blood pressure in pregnant and postpartum patients who are treated with nifedipine and labetalol for severe range blood pressures defined as greater than 160/110. These anti-hypertensives are first line therapy for management of severe range blood pressures in pregnancy and postpartum by the American Congress of Obstetricians and Gynecologist (ACOG).

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients from 20 weeks to up to 6 weeks postpartum
* between the ages of 18-55.
* persistent severe range blood pressures (2 readings or more within 15 minutes) of either 160mmHg systolic or 110mmHg diastolic.

Exclusion Criteria:

* multiple gestation
* patients with non-reassuring fetal heart rate (category 3)
* patients with abruptio placenta
* patients with renal impairment
* history of heart failure
* history of cardiac arrhythmia
* use of anti-hypertensive medications in the past 24 hours
* patients with allergies or medical contraindications to labetalol or nifedipine.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lois Brustman, MD, Study Director — Icahn School of Medicine at Mount Sinai; Howard Minkoff, MD, Study Director — Icahn School of Medicine at Mount Sinai; Poroshat Shekarloo, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Maimonides Hospital, Brooklyn, New York
  - Mount Sinai West, New York, New York

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at two urban academic institutions with participants enrolled from September 2017 to April 2019.
Groups:
- Oral Nifedipine: Oral medication 10mg and 20mg
  Nifedipine: Nifedipine 10mg oral given and the MAP calculated 20 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, nifedipine 20mg oral given and the MAP calculated 20 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, nifedipine 20mg oral given and the MAP calculated 20 minutes after medication is given and institution specific protocol performed.
- Intravenous Labetalol: Intravenous medication 20mg, 40mg, 80 mg
  Labetalol: Labetalol 20mg IV given over 2 minutes and the MAP calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, labetalol 40mg IV given over 2 minutes and the MAP calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, labetalol 80mg IV given over 2 minutes and the MAP calculated 10 minutes after medication is given. If SBP is ≥160mmHg or DBP is ≥110mmHg, then another medication chosen based on institution specific protocol.
Period: Overall Study
Arm/Group | Oral Nifedipine | Intravenous Labetalol
Started | 54 | 55
Completed | 54 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Labetalol | Oral Nifedipine | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.49 (6.25) | 33.67 (5.74) | 34.59 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 20 | 22 | 42
  White, Asian, or Hispanic | 35 | 32 | 67
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.89 (6.36) | 29.84 (6.54) | 28.86 (6.50)
Gestational age [Median (Inter-Quartile Range); unit: weeks] — Population: Data for participants pregnant at baseline
  weeks
    number analyzed (Participants) | 53 | 49 | 102
    (all) | 37.4 [36.3 to 38.6] | 36.9 [34.6 to 38.9] | 37.1 [35 to 38.7]
Number of participants who are Post-partum [Count of Participants; unit: Participants] | 2 | 5 | 7
Number of Participants with Chronic Hypertension (CHTN) [Count of Participants; unit: Participants] | 9 | 9 | 18
Number of Participants with Gestational Hypertension (GHTN) [Count of Participants; unit: Participants] | 12 | 14 | 26
Number of Participants with Diabete Mellitus Type I or II [Count of Participants; unit: Participants] | 2 | 2 | 4
Family History of HTN [Count of Participants; unit: Participants] | 26 | 29 | 55
History of Smoking [Count of Participants; unit: Participants] | 9 | 12 | 21
Pre-medication, Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 173.96 (12.74) | 171.74 (11.19) | 172.86 (11.99)
Pre-medication, DiastolicBlood Pressure [Mean (Standard Deviation); unit: mmHg] | 94.18 (10.02) | 97.09 (10.28) | 95.62 (10.21)

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Non Severe Range Blood Pressure
Description: Time to achieve goal blood pressure, that is, non severe range blood pressures after medication received.
Time Frame: Ten minute intervals from the time of the first severe range blood pressure, up to 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intravenous Labetalol | Oral Nifedipine
Number analyzed (Participants) | 55 | 54
minutes | 10 [10 to 20] | 20 [20 to 30]

2. Primary Outcome: Number of Participants to Achieve Non Severe Range Blood Pressure
Description: Number of participants by ethnicity to achieve goal blood pressure, that is, non severe range blood pressures after medication received.
Time Frame: up to 1 hour
Population: participants by ethnicity
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Labetalol | Oral Nifedipine
Number analyzed (Participants) | 55 | 54
Participants
  White, Asian, and Hispanic: number analyzed (Participants) | 35 | 32
  White, Asian, and Hispanic | 33 | 31
  Black: number analyzed (Participants) | 20 | 22
  Black | 18 | 22

3. Secondary Outcome: Frequency of Genetic Variants of Genes
Description: the frequency of variant alleles in different receptors involved in the response to labetalol and nifedipine administration in the pregnant and postpartum population.
Time Frame: up to 1 year
Population: data not collected
Arm/Group | Intravenous Labetalol | Oral Nifedipine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Medication Side Effects
Description: Number of participants with side effect profile to assess the rate of side effects from IV labetalol and oral nifedipine
Time Frame: assessed 10 minutes to 1 hour after medication is given
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Labetalol | Oral Nifedipine
Number analyzed (Participants) | 55 | 54
Participants
  Headache | 6 | 10
  Nausea | 3 | 7
  Vomiting | 2 | 3
  Dizziness | 8 | 4
  Flushing | 7 | 7
  Any of the above | 18 | 15

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Intravenous Labetalol | Oral Nifedipine
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Labetalol (N=55) | Oral Nifedipine (N=54)
symptomatic hypotenstion (Pregnancy, puerperium and perinatal conditions) | 0 | 1

LIMITATIONS AND CAVEATS:
Small sample size and the study was not double blind

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03506724/Prot_SAP_000.pdf